CLINICAL TRIAL: NCT01999153
Title: Evaluation of the Analgesic Effect of Ropivacaine in Topical Use at the Thin Skin Graft Donor Site
Acronym: ROPI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/119/HP
Record Dates: First submitted 2013-07-29; First posted 2013-12-03 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Graft Pain
Keywords: skin graft; donor site
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRUG : ROPIVACAINE (Experimental): 20 mL topically used during alginate dressing
  Interventions: Drug: 20 mL topically used during alginate dressing NAROPEINE
- PLACEBO : NaCl 0.9 % (Placebo Comparator): 20 mL topically used during alginate dressing
  Interventions: Drug: 20 mL topically used during alginate dressing NaCl

INTERVENTIONS:
Drug: 20 mL topically used during alginate dressing NAROPEINE — 20 mL topically used during alginate dressing
  Other Names: Brand name of drug use NAROPEINE
  Arms: DRUG : ROPIVACAINE
Drug: 20 mL topically used during alginate dressing NaCl — 20 mL topically used during alginate dressing
  Other Names: NaCl 0.9 %
  Arms: PLACEBO : NaCl 0.9 %

SUMMARY:
The aim of the study is to Evaluate of the analgesic effect of ropivacaine in topical use at the thin skin graft donor site.

For Patient needing a thin skin graft < 320 cm2, randomization will be done in 2 groups, one receiving the standard treatment (20 mL of physiologic serum) during the surgical intervention in topical use to recover an alginate dressing (Algosteril)and the other receive 20 mL of Naropein during the surgical intervention on alginate dressing.

The hypothesis of the study is the administration of ropivacaine will decrease the post-operative pain compared to physiologic serum

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patient needing a thin skin graft < 320 cm2 and which is possible on the thigh
* Patient who read the information letter and signed the informed consent
* Patient affiliated at a social security system
* Effective contraceptive method for more than 3 months for women of childbearing age

Exclusion Criteria:

* Contraindication to one of the medicine used (allergy, intolerance, potential drug interaction)
* Treatment by classII or III of analgesics or analgesic dose of aspirin(>500mg per day) at the inclusion or randomization time
* Preoperative EVA>0 at the skin graft donor site on the thigh
* Sensory disturbances of the lower limbs
* Cognitive disturbances not allowing investigations
* Pregnant or lactating women
* People deprived of discernment
* People deprived of their liberty by judicial or administrative authority
* Protected adult (guardianship or trusteeship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-12-09 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Class II analgesic consumption between the 2 arms | 5 days post-operative
  Evaluate the effect of ropivacaine in topical use on an alginate dressing by evaluating the use of class II analgesic medicines in patient who had a thin skin graft

SECONDARY OUTCOMES:
Class II antalgic consumption between the 2 arms | Day 90
  evaluate the effect of ropivacaine on postoperative pain at the skin graft donor site
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | day 90
  potential side effects of ropivacaine on the healing of skin graft donor site

CONTACTS AND LOCATIONS:
Overall Officials: Dorothée COQUEREL-BEGHIN, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- UHRouen, Rouen, France